CLINICAL TRIAL: NCT01936298
Title: Robot-assisted Rehabilitation of Hand by Paralysis of the Upper Limb After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiara Mulé (Other)
Responsible Party: Sponsor-Investigator, Chiara Mulé, Physiatrist Physician, Habilita, Ospedale di Sarnico
Organization: Habilita, Ospedale di Sarnico (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLO01
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Stroke
Keywords: Hand Edema; Exercise Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-ROM Continuous Passive Rehabilitation (Experimental): The group of patients with Active Range Of Motion (A-ROM) is subjected to two session per day in the morning and in the afternoon over a period of two weeks (5 days per week). Each session is composed by 30 min of continuous passive motion rehabilitation and 60 min of physical and occupational therapy.
  Interventions: Device: A-ROM Continuous Passive Rehabilitation
- P-ROM Continuous Passive Rehabilitation (Experimental): The group of patients with Passive Range Of Motion (P-ROM), i.e. without active movements of the hand at the baseline, is subjected to two session per day in the morning and in the afternoon over a period of two weeks (5 days per week). Each session is composed by 30 min of continuous passive motion rehabilitation and 60 min of physical and occupational therapy.
  Interventions: Device: P-ROM Continuous Passive Rehabilitation

INTERVENTIONS:
Device: A-ROM Continuous Passive Rehabilitation — Half an hour of treatment during the morning with the "sequential" program (each finger is mobilized individually) and half an hour of treatment during the afternoon with the "synchronous" program (II-III-IV-V finger are mobilized simultaneously, the thumb individually).
  Other Names: Continuous Passive Motion device for hand: Gloreha
  Arms: A-ROM Continuous Passive Rehabilitation
Device: P-ROM Continuous Passive Rehabilitation — Half an hour of treatment during the morning with the "sequential" program (each finger is mobilized individually) and half an hour of treatment during the afternoon with the "synchronous" program (II-III-IV-V finger are mobilized simultaneously, the thumb individually).
  Other Names: Continuous Passive Motion device for hand: Gloreha
  Arms: P-ROM Continuous Passive Rehabilitation

SUMMARY:
The investigators evaluate the effectiveness of the application of continuous passive motion device for hand rehabilitation in two classes of patients: with a residual active motion and without a residual active motion.

DETAILED DESCRIPTION:
We will conduct a double blind clinical trial. A sample size calculation were performed to determine the necessary number of subjects needed for this study and was based upon the results of a previous pilot study. All patients had functional impairments of their upper extremities after the stroke.

We hypothesized that the hand-rehabilitation oriented with robotics assistance, would improve edema by paralysis of the upper limb even in patient without sensory pathway recovery.

ELIGIBILITY:
Inclusion Criteria:

* a history of acute phase of stroke (less than 12 months post onset),
* first stroke episode,
* no history of peripheral nerve injury or musculoskeletal disease in the affected upper extremity,
* no contracture of the affected wrist or fingers (Modified Ashworth<3),
* no history of any invasive procedure (Botulinum toxin type A) for the treatment of spasticity for at least 6 months before the start of this study,
* for P-ROM patients, the absence of active hand movements,
* for the A-ROM patients, the presence of active hand movements.

Exclusion Criteria:

* unstable medical disorders,
* active Complex Regional Pain Syndrome (CRPS),
* severe spatial neglect,
* aphasia,
* cognitive problems.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Perimeter edema | 1 day after the treatment

SECONDARY OUTCOMES:
Change from Baseline of Visual analogue scale (VAS) | 1 day after the treatment
Change from Baseline of Modified Ashworth Scale for Grading Spasticity (MAS) | 1 day after the treatment
Change from Baseline of Range Of Motion (ROM) | 1 day after the treatment
Clinical Global Impression (CGI) | 1 day after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Mulé, MD, Principal Investigator — Habilita, Ospedale di Sarnico
Locations (1):
- Habilita, Ospedale di Sarnico, Sarnico, Bergamo, Italy

REFERENCES:
- [Background] Yamaguchi T, Tanabe S, Muraoka Y, Imai S, Masakado Y, Hase K, Kimura A, Liu M. Effects of integrated volitional control electrical stimulation (IVES) on upper extremity function in chronic stroke. Keio J Med. 2011;60(3):90-5. doi: 10.2302/kjm.60.90. PMID 21964036
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Kim EH, Chang MC, Seo JP, Jang SH, Song JC, Jo HM. The effect of a hand-stretching device during the management of spasticity in chronic hemiparetic stroke patients. Ann Rehabil Med. 2013 Apr;37(2):235-40. doi: 10.5535/arm.2013.37.2.235. Epub 2013 Apr 30. PMID 23705119
- [Background] Fugl-Meyer AR. Post-stroke hemiplegia assessment of physical properties. Scand J Rehabil Med Suppl. 1980;7:85-93. No abstract available. PMID 6932734
- [Background] Bell A, Muller M. Effects of kinesio tape to reduce hand edema in acute stroke. Top Stroke Rehabil. 2013 May-Jun;20(3):283-8. doi: 10.1310/tsr2003-283. PMID 23841976
- [Background] Bialosky JE, George SZ, Bishop MD. How spinal manipulative therapy works: why ask why? J Orthop Sports Phys Ther. 2008 Jun;38(6):293-5. doi: 10.2519/jospt.2008.0118. Epub 2008 May 27. No abstract available. PMID 18515964
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Kong KH, Chua KS, Lee J. Symptomatic upper limb spasticity in patients with chronic stroke attending a rehabilitation clinic: frequency, clinical correlates and predictors. J Rehabil Med. 2010 May;42(5):453-7. doi: 10.2340/16501977-0545. PMID 20544156
- [Background] Lundstrom E, Smits A, Terent A, Borg J. Time-course and determinants of spasticity during the first six months following first-ever stroke. J Rehabil Med. 2010 Apr;42(4):296-301. doi: 10.2340/16501977-0509. PMID 20461330
- [Background] Villafane JH, Valdes K. Combined thumb abduction and index finger extension strength: a comparison of older adults with and without thumb carpometacarpal osteoarthritis. J Manipulative Physiol Ther. 2013 May;36(4):238-44. doi: 10.1016/j.jmpt.2013.05.004. Epub 2013 May 27. PMID 23719517
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Chang CW, Kuo LC, Cheng YT, Su FC, Jou IM, Sun YN. Reliable model-based kinematics analysis system for articulated fingers. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:4675-8. doi: 10.1109/IEMBS.2007.4353383. PMID 18003049
- [Derived] Borboni A, Villafane JH, Mulle C, Valdes K, Faglia R, Taveggia G, Negrini S. Robot-Assisted Rehabilitation of Hand Paralysis After Stroke Reduces Wrist Edema and Pain: A Prospective Clinical Trial. J Manipulative Physiol Ther. 2017 Jan;40(1):21-30. doi: 10.1016/j.jmpt.2016.10.003. Epub 2016 Nov 12. PMID 27847124